CLINICAL TRIAL: NCT05956223
Title: The Development of a System for Measurement of Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Bionics Institute of Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-1562H; NCT06386822 (obsolete NCT alias)
Record Dates: First submitted 2023-05-22; First posted 2023-07-21 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Essential Tremor; Dystonia
Keywords: Essential Tremor; Dystonia; Virtual Reality; Biokin
MeSH Terms: conditions — Essential Tremor; Dystonia

STUDY DESIGN:
Intervention Model Description: Single group assignment. Up to 90 participants with Essential Tremor and up to 30 Control participants will be recruited to the study. Both groups will undergo the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Virtual Reality & Movement Monitoring (Experimental): Participants will don the equipment used to measure their tremor and replicate a series of standardized movements to measure their tremor, in and out of the VR platform.
  Interventions: Device: Virtual Reality measurement of essential tremor and dystonia

INTERVENTIONS:
Device: Virtual Reality measurement of essential tremor and dystonia — 1. The virtual reality (VR) platform, which detects whole-of-body movements. The VR environment is a series of sensors in a room that detect whole body motion and a series of sensors worn by the participant. As well the participant dons VR "goggles" that allows them to "see" a virtual environment in which they can perform the TETRAS.
     Within the VR platform, an avatar (an electronic image that represents the participant) is produced in the VR environment, and this will be used to review the participant.
  2. Sensors for the detection of wrist, head and voice tremor. The sensors are small devices worn on the wrists and head of the participant and are similar to those used in the VR system. A microphone is attached to the participants to detect voice tremor.

SUMMARY:
The goal of this clinical trial is to develop a system which can be used to measure movements in people with Essential Tremor (with or without dystonia).

The main questions it aims to answer are:

* Can individuals with Essential Tremor be distinguished from individuals without tremor using Virtual Reality (VR)
* Can the current Essential Tremor Assessment Scale (the TETRAS) be reproduced in VR
* Can Essential Tremor be quantified using a measurement system
* Can Dystonia be quantified using a measurement system. Participants will don the equipment used to measure their tremor and replicate a series of standardized movements to measure their tremor, in and out of the VR platform. The assessment will take no longer than an hour.

DETAILED DESCRIPTION:
This study aims to develop a way of objectively measuring the neurological disorders, Essential Tremor (ET) and dystonia. These conditions can affect the upper and lower limbs, head, voice, face and trunk. ET and dystonia can be difficult to assess and treat, particularly if severe, and therapies are limited.

Currently the severity of these conditions is formally assessed by clinician rated scales such as the Essential Tremor Rating Assessment Scale (TETRAS) which is biased towards the upper limbs, requires training and is not objective. There is a need for a more precise, less variable measure of tremor that can used easily be non-expert clinicians. This study questions whether it is possible to quantify ET and dystonia using a measurement system in a virtual reality (VR) environment.

Data will be collected from measurement sensors embedded in the VR environment from healthy control participants, and those with ET with and without dystonia. Participants will be placed in a VR environment and instructed to perform the TETRAS. This will help to develop an algorithm which can measure ET severity using machine learning. It is expected that the algorithm will provide a better assessment of ET and dystonia than the TETRAS. This study may pave the way towards the development of simpler devices to which the algorithm can be applied.

ELIGIBILITY:
Inclusion Criteria - Control participants

* Aged 18 to 80 years
* Able to provide informed consent for self
* Able to comply with all study procedures

Exclusion Criteria -Control participants

* Any neurological disorder
* Any other non-neurological cause of tremor e.g. medication induced

Inclusion Criteria - ET participants

* Aged 18 to 80 years
* Able to provide informed consent for self
* Clinical diagnosis of ET or ET plus syndrome
* Able to comply with all study procedures

Exclusion Criteria - ET Participants

* Tremor other than ET (e.g. parkinsonian, functional tremor)
* Presence of other movement disorder
* For Deep Brain Stimulation (DBS) participants: unwilling or unable to turn off and on their own stimulator for the duration of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
1. To quantify Essential Tremor and dystonia using a measurement system | At enrolment. This study is a single assessment conducted at one time point.
  Using commercially available Virtual Reality (VR) equipment and a commercially available Inertial Measurement Unit (IMU), the presence of the tremor and dystonia in participants with Essential Tremor will be measured and their severity rated.

CONTACTS AND LOCATIONS:
Overall Officials: David Szmulewicz, MBBS PhD, Principal Investigator — The Royal Victorian Eye and Ear Hospital
Locations (1):
- The Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
None. No findings of direct clinical relevance are expected.